CLINICAL TRIAL: NCT06294119
Title: Multivariate Approach to the Numerical Assessment of Cortical - Autonomic - VAscular Dynamic Interplay
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Policlinico S. Donato (Other)
Responsible Party: Principal Investigator, Marco Ranucci, Principal Investigator, IRCCS Policlinico S. Donato
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MANCAVA; 2022SLB5MX (Other Grant/Funding Number: Italian Ministry of Research)
Record Dates: First submitted 2024-02-27; First posted 2024-03-05 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Cardiac Disease; Depression
MeSH Terms: conditions — Heart Diseases; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cardiac surgery (Other): An experimental setup will be devised for the simultaneous monitoring and recording of EEG, ECG, AP, and R together with CBF in patients scheduled for major cardiac surgery. Recording sessions will take place 1 day before (PRE) and within 7 days after (POST) surgery. The experimental protocol including physiological data recordings includes three sessions lasting 10 minutes each: a session at resting state in supine position, a session during autonomic challenge obtained via active standing evoking reflex sympathetic activation, and a session of emotional elicitation via the administration of videos. The overall duration of the experiment is therefore 30 minutes in PRE and POST. A total of 40 short video clips of the duration of 15 seconds each will be presented to a total of 80 voluteers will be recruited for the MANCAVA study.
  Interventions: Procedure: Major Cardiac surgery

INTERVENTIONS:
Procedure: Major Cardiac surgery — From a clinical perspective, MANCAVA will especially target neuro-cardiovascular health and mood disorders such as depression

SUMMARY:
MANCAVA sets out fundamental methodologies for characterizing human fundamental physiological system interactions at a whole-body level, particularly focusing on the interplay among cortical brain activity, autonomic function, and cerebrovascular autoregulatory mechanisms. By investigating the complex, time-varying mechanisms underlying the multisystem dynamic interactions, novel methods linking various brain areas and reflex functions to target organs and districts such as heart and circulatory system are proposed with the clinical aim linked to the emerging topic of depression.

In this scenario, proper new mathematical tools will allow a significant leap from the current state of the art, paving the way towards a new understanding of leading comorbid contributors to global diseases such as cardiac and cerebrovascular morbidity in mood disorders. In turn, this will provide an integration among physiological and psychological dimensions for a more holistic view on depression.

Researchers, professionals, and patients will all benefit from a comprehensive assessment of brain-mind-body interplay, leading to the new extended definition of default mode/mood network, neurovascular-evoked responses to autonomic stimuli, brain-autonomic consequences of emotional responses, and physiological substrates of depressive states.

ELIGIBILITY:
Inclusion Criteria:

* age older than 18 years
* spontaneous sinus rhythm
* signed informed consent
* indication to heart surgery

Exclusion Criteria:

* age lower than 18 years
* absence of sinus rhythm
* pregnancy
* impossibility of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-05-08 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Autoregulation index (ARI) | 24 months
  ARI is an index describing the state of cerebral autoregulation from mean cerebral blood velocity and mean arterial pressure. It ranges between 1 and 9. ARI>4 means working autoregulation. ARI<4 means impaired autoregulation. It will be computed for all participants in PRE and POST.
number of patients developing depression | 24 months
  The number of patients developing depression will be assessed by the results of psychometric tests
Baroreflex sensitivity | 24 months
  Baroreflex sensitivity will be measured in ms/mmHg. A higher value means a better baroreflex regulation. It will be computed in all participants in PRE and POST surgery.
Cortical activity | 24 months
  Power of EEG in Alpha and Beta band will be measured in square microvolt

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Policlinico San Donato, San Donato Milanese, Milan, Italy

IPD SHARING:
Plan to Share IPD: No